CLINICAL TRIAL: NCT05644496
Title: A Randomized Controlled Trial of ZYNRELEF Versus Standard of Care for Pain Management Following Unilateral Total Knee Arthroplasty
Brief Title: ZYNRELEF for Pain Management in Total Knee Arthroplasty
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Baptist Health South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1891382
Record Dates: First submitted 2022-11-11; First posted 2022-12-09 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Post Operative Pain; Osteoarthritis, Knee
Keywords: Knee Arthroplasty; Postoperative pain management
MeSH Terms: conditions — Pain, Postoperative; Osteoarthritis, Knee | interventions — bupivacaine-meloxicam drug combination

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intervention (Experimental): In addition to the standard-of-care arm description, single administration of Bupivacaine-Meloxicam 400 Mg-12 Mg/14 mL Injectable Solution, Extended Release in the surgical site before complete wound closure.
  Interventions: Drug: Bupivacaine-Meloxicam 400 Mg-12 Mg/14 mL Injectable Solution, Extended Release
- Standard-of-care (No Intervention): Usual standard of care procedure for knee replacement and pain management before, during and immediately following surgery.

INTERVENTIONS:
Drug: Bupivacaine-Meloxicam 400 Mg-12 Mg/14 mL Injectable Solution, Extended Release — Instillation of the drug into the knee joint capsule and surrounding tissues after placing the knee prosthesis and before close of the surgical wound
  Other Names: Zynrelef
  Arms: Intervention

SUMMARY:
The goal of this randomized controlled trial is to compare opioid medication consumption after surgery for patients who have a total knee replacement.

The main questions it aims to answer are:

* How well does the study drug control pain in the days after surgery?
* Does the study drug reduce the amount of opioid analgesic consumed after surgery?

Participants in the study group will undergo a total knee replacement as planned with their surgeon. In addition, be given the study drug, Zynrelef (combination of bupivacaine and meloxicam).

Researchers will compare the above to a control group who will have a total knee replace only according to usual standards to see if there are any differences in the amount of a type of pain medication (opioid analgesic) consumed in the days following surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients undergoing primary unilateral total knee arthroplasty [Current Procedural Terminology Code: 27447]
2. Patients with a diagnosis of primary osteoarthritis [ICD-10 codes: M17.0, M17.10, M17.11, M17.12]
3. Varus deformity less than 10 degrees
4. Flexion contracture less than 10 degrees
5. Age 35 - 70 years old
6. BMI < 40
7. Patients who are discharged on the same day after the unilateral total knee arthroplasty procedure

Exclusion Criteria:

1. Inflammatory arthritis
2. Post-traumatic arthritis
3. Valgus deformity
4. Severe varus (> 10 degrees)
5. Severe flexion contracture (> 10 degrees)
6. Overnight or longer hospital stay after surgery
7. Prior surgery on affected knee other than knee arthroscopy for meniscal or cartilage debridement/repair
8. Creatinine > 1.2
9. Chronic Kidney Disease (CKD) stage 3, 4, 5 or end stage renal disease
10. Uncontrolled Diabetes mellitus (Glycated Hemoglobin > 8.0%)
11. Current liver disease
12. Personal history of depression or anxiety disorder
13. Personal history of Deep Venous Thrombosis (DVT) or Pulmonary Embolism (PE)
14. Narcotic or tramadol use within 2 weeks of the planned procedure
15. Allergy to aspirin, NSAIDS, oxycodone, Tylenol, local anesthetics
16. Walking aid for anything other than the operative joint
17. Contraindication for use of the study drug (as specified by the manufacturer):

    * Known hypersensitivity to local amide anesthetics, NSAIDs or study drug components
    * History of asthma, urticaria or other allergic-type reactions to aspirin or other NSAIDs
18. Patients taking the following medications:

    * Amitriptyline
    * Nortriptyline
    * Gabapentin
    * Pregabalin
    * Duloxetine (SNRI)
    * Des-Venlafaxine (SNRI)
    * Cyclobenzaprine
    * Baclofen
19. Pregnant or lactating females
20. Patients unable to provide informed consent
21. Subjects who, in the opinion of the Investigator, may be non-compliant with study schedules or procedures

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Estimated)
Dates: Start 2023-03-09 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Total opioid analgesic consumption | 5 days following surgical procedure
  Amount of opioid analgesic consumed in the time frame calculated as Morphine Milligram Equivalent (MME).
Change in pain assessment scores | Baseline and every 24 hours for 120 hours following surgical procedure
  Pain assessment scores using the pain Numeric Rating Scale for pain (NRS).
  The NRS scale is measured on a scale of 0 - 10, where 0 is no pain and 10 is the most severe pain.

SECONDARY OUTCOMES:
Incidence of major complications | 42 days following surgical procedure
  Number of procedure-related adverse events and medication-related adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Juan C Suarez, MD, Principal Investigator — Baptist Health South Florida
Locations (1):
- Doctors Hospital, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No